CLINICAL TRIAL: NCT00196196
Title: A Precision and Accuracy Study of the Codman Valve Position Verification (VPV) System.
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Codman & Shurtleff (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VPV-US03-001
Record Dates: First submitted 2005-09-12; First posted 2005-09-20 (Estimated); Results first posted 2008-12-05 (Estimated); Last update posted 2012-05-28 (Estimated); Status verified 2011-02

CONDITIONS: Hydrocephalus; Normal Pressure Hydrocephalus
Keywords: Hydrocephalus; Codman Hakim Programmable Valve; Programmable Valve; Shunt System
MeSH Terms: conditions — Hydrocephalus; Hydrocephalus, Normal Pressure

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Codman VPV System — Valve Positioning Verification (VPV) System

SUMMARY:
The purpose of this study is to determine the agreement rate between the CODMAN Valve Position Verification (VPV) adjustment outcome (reprogramming) and X-ray verification in order to support an alternative to X-ray confirmation with respect to the valve adjustment process.

DETAILED DESCRIPTION:
Patients with Hydrocephalus, managed with an implanted Codman HakimTM Programmable Valve (CHPV), occasionally visit their physician to have their valve adjusted to a different setting to manage their condition. After the adjustment, an x-ray of the skull is taken to confirm the valve setting.

The Codman VPV System is designed to facilitate and confirm the adjustment of a CHPV. After signing the informed consent, Subjects will be enrolled in the study and have their CHPV adjusted using the Codman VPV System. After the adjustment, an x-ray of the skull will be taken to verify the valve setting. No further follow up visit is needed after the adjustment.

This study is expected to enroll about 300 Subjects from up to 20 sites in the United States.

ELIGIBILITY:
Inclusion Criteria:

* A CODMAN Hakim Programmable Valve (CHPV) has been implanted for the management of the Subject's Hydrocephalus.
* The Subject has given written informed consent prior to enrolling in the study.
* The Subject requires adjustment of the CODMAN Hakim Programmable Valve (CHPV) for the management of Hydrocephalus·
* The Subject's implanted CHPV will be adjusted using the Implanted Valve Mode.

Exclusion Criteria:

* The Subject's valve is located in the deep lumbar position.
* The Subject has an open and/or recent wound site in the region of the implanted valve.
* The Subject has a history of Ultrasound gel allergies.
* The Subject is a prisoner.
* The subject has been previously enrolled in this protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 274 (Actual)
Dates: Start 2004-09; Primary Completion 2006-10 (Actual); Study Completion 2006-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: J. Thomas Megerian, MD, Study Director — Codman & Shurtleff
Locations (8):
- United States (8):
  - Phoenix, Arizona
  - Orlando, Florida
  - Boston, Massachusetts
  - Newark, New Jersey
  - New York, New York
  - Cleveland, Ohio
  - Portland, Oregon
  - Richardson, Texas

REFERENCES:
- [Background] Bret P, Guyotat J, Ricci AC, Mottolese C, Jouanneau E. [Clinical experience with the Sp[hy adjustable valve in the treatment of adult hydrocephalus. A series of 147 cases]. Neurochirurgie. 1999 May;45(2):98-108; discussion 108-9. French. PMID 10448649
- [Background] Petrie A, Sabin C. Medical Statistics at a Glance. Blackwell Science Ltd: 90-91
- [Background] American Society of Radiologic Technologists, Statement on IOM Report, "To Err Is Human: Building a Safer Health System", www.asrt.org/other_categories/government_relations/iom_report.htm
- [Background] Pollack IF, Albright AL, Adelson PD. A randomized, controlled study of a programmable shunt valve versus a conventional valve for patients with hydrocephalus. Hakim-Medos Investigator Group. Neurosurgery. 1999 Dec;45(6):1399-408; discussion 1408-11. doi: 10.1097/00006123-199912000-00026. PMID 10598708
- [Background] Rohde V, Mayfrank L, Ramakers VT, Gilsbach JM. Four-year experience with the routine use of the programmable Hakim valve in the management of children with hydrocephalus. Acta Neurochir (Wien). 1998;140(11):1127-34. doi: 10.1007/s007010050226. PMID 9870057
- [Background] Zemack G, Romner B. Seven years of clinical experience with the programmable Codman Hakim valve: a retrospective study of 583 patients. J Neurosurg. 2000 Jun;92(6):941-8. doi: 10.3171/jns.2000.92.6.0941. PMID 10839253

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Subjects were enrolled between September 29, 2004 and October 13, 2006. Twelve (12) investigational sites within the US enrolled 274 Subjects.
Pre-assignment Details: Of the 274 Subjects enrolled, 5 were determined to be ineligible - did not have hydrocephalus, a required condition per inclusion/exclusion criteria. Two (2) Subjects withdrew early. Overall, 267 Subjects were eligible for analysis.
Period: Overall Study
Arm/Group | Codman VPV System
Started | 274
Completed | 267
Not Completed | 7
Not completed — Withdrawal by Subject | 2
Not completed — Did not have required condition (hydroce | 5

BASELINE CHARACTERISTICS:
Arm/Group | Codman VPV System
Number analyzed (Participants) | 267
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 35
  Between 18 and 65 years | 90
  >=65 years | 142
Age Continuous [Mean (Standard Deviation); unit: years] | 57 (26.1)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 137
  Male | 130
Region of Enrollment [Number; unit: participants]
  United States | 267

OUTCOME MEASURES:

1. Primary Outcome: Percentage of Participants Who Achieved "Adjustment Complete" and a Consensus X-ray Reading
Description: Up to 5 attempts to achieve "Adjustment Complete" using the Codman Valve Position Verification (VPV) system for each Subject. Agreement in 2 of 3 valve X-ray readings by independent radiologists for each Subject was considered "consensus X-ray". All participants included achieved "Adjustment Complete" and a "consensus X-ray reading".
Time Frame: Day 1
Measure: Number; unit: Percentage of participants
Arm/Group | Codman VPV System
Number analyzed (Participants) | 267
Percentage of participants | 98.33

2. Secondary Outcome: Percentage of Agreement Between the Codman Valve Position Verification (VPV) System and Consensus X-rays Using Various Thresholds
Description: Percentage of agreement between consensus X-ray readings and the intended setting programmed by the Codman Valve Position Verification (VPV) system. This was assessed at various steps (intervals of mmH20) as increments allow on the Codman Hakim Programmable Valve. (1 step = 10 mmH20, 2 steps = 20 mmH20, +2 steps = >20 mmH20)
Time Frame: Day 1
Measure: Number; unit: Percentage of agreement
Arm/Group | Codman VPV System
Number analyzed (Participants) | 267
Percentage of agreement
  Percentage of Agreement (exact match) | 63.89
  Percentage of Agreement in 1 step (+/- 10 mmH20) | 96.11
  Percentage of Agreement >2 steps (>20 mmH20) | 1.67

ADVERSE EVENTS:
Arm/Group | Codman VPV System
Serious Adverse Events (participants affected / at risk) | 0/0
Other Adverse Events (participants affected / at risk) | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: embargo of 60 days or less